CLINICAL TRIAL: NCT02295761
Title: Promoting Overweight Adolescents Physical Activity and Adherence to Healthy Lifestyles: a Randomized Controlled Trial
Brief Title: Promoting Overweight Adolescents Physical Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heidi Ruotsalainen (Other)
Responsible Party: Sponsor-Investigator, Heidi Ruotsalainen, researcher, University of Oulu
Organization: University of Oulu (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 100/2011
Record Dates: First submitted 2014-02-18; First posted 2014-11-20 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
Keywords: motor activity; obesity; overweight; intervention study; health promotion; lifestyle counseling; adherence
MeSH Terms: conditions — Obesity; Motor Activity; Overweight | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Active Comparator): 12-weeks
  Interventions: Behavioral: Lifestyle counseling (Fb)
- Lifestyle counseling + activity watch (Active Comparator): 12-weeks
  Interventions: Behavioral: Lifestyle counseling + activity monitor (Fb+Act)

INTERVENTIONS:
Behavioral: Lifestyle counseling (Fb) — Facebook-delivered lifestyle counseling
  Arms: Lifestyle counseling
Behavioral: Lifestyle counseling + activity monitor (Fb+Act) — Facebook-delivered lifestyle counseling and self-monitoring physical activity using Polar activity monitor
  Arms: Lifestyle counseling + activity watch

SUMMARY:
Objectives: Aim of this study is to evaluate the effectiveness of Facebook-delivered lifestyle counseling intervention on overweight and obese adolescent's physical activity, BMI and adherence to healthy lifestyles.

Design: A 12-week, randomized controlled trial with three, 24 and 36 month follow-up.

Settings: One of the Northern Finland healthcare districts school health care units.

Participants: all overweight or obese 13-16 years old adolescent and their parents were invited to study.

Methods: Adolescents were stratified by gender, age, and self-reported physical activity and they were randomized into three groups. Two experimental groups, where those both got Facebook-delivered lifestyle counseling and one of the experimental groups got activity monitor which showed the daily activity. One group served as a control group. Parents were allocated to intervention groups according which group their adolescent were randomized.

Outcomes: physical activity,body mass index (BMI) adherence to healthy lifestyles. Baseline measurements have been done and assessment to adherence to healthy lifestyles have been measured. Follow-up measures have been conducted three months after baseline. Adherence to healthy lifestyles measurement follow-up is at 24 and 36 months after intervention.

DETAILED DESCRIPTION:
Adolescents inclusion criteria: weight-fof-height over 20% over normality (finnish recommendations), age 13-16 years old Exclusion criteria: mental health problems, or long term illness.

Adolescents outcome measures:

1. Change from baseline physical activity at 12 weeks using a blinded Polar Activity activity monitor. Primary outcome is measuder using continuous scale and measurement unit is one minute. For each subject the minutes per day is calculated (minimum value is 0).

   It is a wrist worn uni-axial accelerometer designed to determine physical activity of children and adolescents. Polar activity monitor records activity in every 30 seconds bouts and the device records steps when user takes >70 steps per minute. Activity measurements were done for 21 days at baseline and three months follow-up measurements. A wear-time shows valid days in this study, and one valid day required at least 500 minutes / day and users had to have at least eight valid days from weekdays and also one from weekend.

   The device integrates the total amount of acceleration in one dimension and counts physical activity quantity and quality, amount of steps and total energy expenditure in calories (Kcal). Physical activity is defined by metabolic equivalent of tasks (MET), which are divided in five areas of activity; very light (1-2 MET), light (2-3.5 MET), moderate (3.6-5 MET), vigorous (5.1-8 MET) and vigorous plus (>8 MET).
2. Change from baseline body mass index (BMI) at 12 weeks BMI was calculated from weight (kg) and height (cm) that were measured by heath care professionals. Formula BMI= weight (kg)/(height (m))2 were using calculating BMI. Scale is continuous.
3. Change from baseline adherence to healthy lifestyles at 12 weeks, 24 months and 36 months. The Adherence to healthy lifestyle is measured using Likert scale with 5 point. The range were from 1 to 5, where 1=strong disagree - 5=strong agree. The adherence to healthy lifestyle questionnaires validity and reliability have been tested before (Kyngäs et al. 2000. The development of an instrument to measure the compliance of adolescents with a chronic diseases. Journal of advanced nursing 32 (6):1499-1506.

Parents outcomes:

1) Change from baseline adherence to healthy lifestyles at 12 weeks, 24 months and 36 months. The Adherence to healthy lifestyle is measured using Likert scale with 5 point. The range were from 1 to 5, where 1=strong disagree - 5=strong agree. The adherence to healthy lifestyle questionnaires validity and reliability have been tested before (Kyngäs et al. 2000. The development of an instrument to measure the compliance of adolescents with a chronic diseases. Journal of advanced nursing 32 (6):1499-1506.

Data analysis: Across-group comparison of baseline physical activity, BMI, gender and age were conducted for evaluable participants using ANOVA (Kruskal-Wallis test) for continuous variables and for categorical variables (eg. sex) we used Fischer´s exact test.

ELIGIBILITY:
Inclusion Criteria:

* 13-16 years old,
* overweight or obese (weight for height >20% over normality)

Exclusion Criteria:

* mental health problems, long term illnesses.

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline physical activity at 12 weeks | 12 weeks
  Adolescent primary outcome is measuder using continuous scale and measurement unit is one minute.
  It is a wrist worn uni-axial accelerometer designed to determine physical activity of children and adolescents. Polar activity monitor records activity in every 30 seconds bouts and the device records steps when user takes >70 steps per minute. Activity measurements were done for 21 days at baseline and three months follow-up measurements. A wear-time shows valid days in this study, and one valid day required at least 500 minutes / day and users had to have at least eight valid days from weekdays and also one from weekend.

SECONDARY OUTCOMES:
Change from baseline adherence to healthy lifestyle at 12 weeks, 24 and 36 months | 12 weeks, 24 and 36 months
  adolescent secondary outcome, parents primary outcome. The Adherence to healthy lifestyle is measured using Likert scale with 5 point. The range were from 1 to 5, where 1=strong disagree - 5=strong agree. The adherence to healthy lifestyle questionnaires validity and reliability have been tested before (Kyngäs et al. 2000. The development of an instrument to measure the compliance of adolescents with a chronic diseases. Journal of advanced nursing 32 (6):1499-1506.
Change from baselin BMI at 12 weeks | 12 weeks
  adolescent secondary outcome BMI is calculated from weight (kg) and height (cm) that were measured by heath care professionals. Formula BMI= weight (kg)/(height (m))2 were using calculating BMI. Scale is continuous.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi M Ruotsalainen, MHS, Principal Investigator — University of Oulu, institute of Health sciences
Locations (1):
- University of Oulu, institute of health sciences, Oulu, Finland

REFERENCES:
- [Derived] Ruotsalainen H, Kyngas H, Tammelin T, Heikkinen H, Kaariainen M. Effectiveness of Facebook-Delivered Lifestyle Counselling and Physical Activity Self-Monitoring on Physical Activity and Body Mass Index in Overweight and Obese Adolescents: A Randomized Controlled Trial. Nurs Res Pract. 2015;2015:159205. doi: 10.1155/2015/159205. Epub 2015 Dec 1. PMID 26697218